CLINICAL TRIAL: NCT07153900
Title: Safety Evaluation of BACK4 Device
Brief Title: BACK4 Safety Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWIMS America Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF-B4-001
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Safety and Tolerability in Healthy Subjects
Keywords: muscle stimulation; topical heating
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hands-on (Active Comparator): Treatment delivered by therapist utilizing multipolar electrode
  Interventions: Device: Treatment with BACK4 System
- Hands-free (Active Comparator): Treatment delivered utilizing fixed pads
  Interventions: Device: Treatment with BACK4 System

INTERVENTIONS:
Device: Treatment with BACK4 System — Use of combined RF and EMS therapy with BACK4 Device

SUMMARY:
To characterize the safety of combined RF and EMS therapies with the BACK4 device in healthy volunteers. Subjects will receive 3 treatments of increasing intensity over a one week period.

ELIGIBILITY:
Inclusion Criteria:

* Adults 22-55 years old
* Able to provide written informed consent

Exclusion Criteria:

* Injury within the past 30 days
* Cancer or cancerous lesions in the treatment area
* Skin disorders (e.g., eczema, shingles), skin burns, or open wounds
* Coagulation disorders, phlebitis, or thrombophlebitis
* Insensitivity to heat
* Local insensitivity to pain and/or touch
* Fever, bacterial infection, infectious disease, or tuberculosis
* Severe hypertension or hypotension
* Electrical implants (e.g., pacemaker, insulin pump, neurostimulator)
* History of seizures or recent surgery
* Known hypersensitivity to device materials
* Pregnant or breastfeeding women
* Participation in another clinical trial within 30 days

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with a reported Adverse Event | 7 days
  Characterize the number of adverse events for the combined use of RF and EMS with the BACK4 device across the device's intended configurations

SECONDARY OUTCOMES:
Number of participants with a device-related adverse event | 7 days
  Characterize the number of device-related adverse events for the combined use of RF and EMS in terms of with the BACK4 device across the device's intended configurations
Number of patients reporting therapy tolerability | 7 days
  Therapy tolerability assessment will be ascertained by the subject using a 5-point scale (1=very uncomfortable, 2=somewhat uncomfortable, 3=neutral, 4=somewhat comfortable, 5=very comfortable)

CONTACTS AND LOCATIONS:
Locations (1):
- RORE Method, Birmingham, Michigan, United States

IPD SHARING:
Plan to Share IPD: No